CLINICAL TRIAL: NCT07310810
Title: Mulligan Mobilization Versus Extracorporeal Shockwave Therapy on Ultrasonographic Changes in Patients With Adhesive Capsulitis
Brief Title: Mulligan Mobilization vs Shockwave Therapy in Adhesive Capsulitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ragab Gaber, lecturer assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 012/005863
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Adhesive Capsulitis
Keywords: Adhesive capsulitis; Mulligan mobilization; EXTRACORPOREAL SHOCKWAVE THERAPY; ULTRASONOGRAPHIC CHANGES
MeSH Terms: conditions — Bursitis | interventions — Movement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- - Group A (study group) (Experimental): received mulligan technique and conventional treatment
  Interventions: Other: Mulligan mobilization; Other: Conventional treatment
- Group B (study group) (Experimental): received extracorporeal shockwave therapy and conventional treatment.
  Interventions: Device: Shockwave; Other: Conventional treatment
- Group C (control group) (Experimental): received conventional treatment only.
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Device: Shockwave — From sitting with shoulder abducted at 45 degree and elbow flexed and the forearm rested on flat surface, The patients in the intervention group B received shock wave therapy once a week for 4 weeks. The focus probe sets were used and, in each session, patients received ESWT from anterior and posterior directions (on the average 1200 shocks between 0.1 and 0.3 mJ/mm2) up to the maximum threshold of pain tolerance in the shoulder
  Arms: Group B (study group)
Other: Mulligan mobilization — Mobilization with movement (MWM) is the concurrent application of sustained accessory mobilization applied by a therapist and an active physiological movement to end range applied by the patient. Passive end-of-range overpressure, or stretching, is then delivered without pain as a barrier
  Other Names: Mobilization with movement
  Arms: - Group A (study group)
Other: Conventional treatment — Conventional treatment will be axillary ultrasound and laser ,low loading stretching exercise and home program exercises

SUMMARY:
To investigate and compare the effects of Mulligan mobilization versus shock wave therapy in patients with adhesive capsulitis on Pain intensity level, Range of motion, Functional disability level, Ultrasonographic changes (soft tissue thickness) and Hand grip strength.

DETAILED DESCRIPTION:
sixty patients of both genders according to sample size calculation, referred from orthopedist, diagnosed adhesive capsulitis patients. they screened according to inclusion and exclusion criteria. Their age between 40 and 60 years was randomly allocated to three treatment groups.

* Group A (study group) (n=20) will receive mulligan technique and conventional treatment.
* Group B (study group) (n=20) will receive extracorporeal shockwave therapy and conventional treatment.
* Group C (control group) (n=20) will receive conventional treatment only.

Inclusion criteria: patients that will be included in the study will be referred from orthopedic physician with:

1. Patients referred from orthopedist and diagnosed as frozen shoulder
2. The age of the participant will be from 40-60 (Agarwal S., et al.2016).
3. Body mass index from 25- 30 kg/m2.
4. having a painful stiff shoulder for at least 3 months
5. having limited ROM of a shoulder joint (ROM losses of 25% or greater compared with the noninvolved shoulder in at least 2 of the following shoulder motions: glenohumeral flexion, abduction and lateral rotation.
6. ability to complete Disabilities of the Arm, Shoulder and Hand questionnaires (DASH).

Exclusion criteria:

1. history of surgery on the particular shoulder
2. Rheumatoid arthritis
3. painful stiff shoulder after a severe trauma
4. fracture of the shoulder complex
5. rotator cuff rupture
6. tendon calcification.

ELIGIBILITY:
Inclusion Criteria:

Patients referred from orthopedist and diagnosed as frozen shoulder The age of the participant will be from 40-60 (Agarwal S., et al.2016). Body mass index from 25- 30 kg/m2. having a painful stiff shoulder for at least 3 months having limited ROM of a shoulder joint (ROM losses of 25% or greater compared with the noninvolved shoulder in at least 2 of the following shoulder motions: glenohumeral flexion, abduction and lateral rotation.

ability to complete Disabilities of the Arm, Shoulder and Hand questionnaires (DASH).

Exclusion Criteria:

history of surgery on the particular shoulder Rheumatoid arthritis painful stiff shoulder after a severe trauma fracture of the shoulder complex rotator cuff rupture tendon calcification.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity level. | 4 weeks
  measured by Visual analog scale
Range of motion. | 4 weeks
  measured by digital goniometer
Functional disability level. | 4 weeks
  Determined by Disabilities of the arm, shoulder and hand questionnaire (DASH)
Soft tissue thickness (Capsule thickness) | 4 weeks
  measured by musculoskeletal ultrasonography
Hand grip strength | 4 weeks
  Measured by hand dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed R Gaber, Asst. lect., Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No